CLINICAL TRIAL: NCT06971250
Title: Peripheral KV7 Activation for Pain Relief - A Randomized, Placebo-Controlled Crossover Microdosing Trial Using Flupirtine
Brief Title: Peripheral KV7 Activation for Pain Relief
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stefan Heber (Other)
Responsible Party: Sponsor-Investigator, Stefan Heber, Principal investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: EK1385/2024
Record Dates: First submitted 2025-05-03; First posted 2025-05-14 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Pain
Keywords: KV7 potassium channels; Flupirtine; Pain modulation; Peripheral analgesia; Experimental pain model; Capsaicin; Microdosing; non-opioid pain treatment; heat pain
MeSH Terms: conditions — Pain | interventions — Capsaicin; flupirtine

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, placebo-controlled, single-visit crossover design in healthy volunteers. Each participant receives multiple intradermal injections in a predefined sequence, with each injection acting as its own control. A balanced Williams design ensures equal distribution of intervention order. The interventions include capsaicin with or without Flupirtine (multiple doses) and heated fluid injections with or without Flupirtine. Pain intensity is measured every 5 seconds using numeric rating scales. The model is optimized for within-subject comparisons of localized, short-duration nociceptive responses and permits precise analysis of peripheral analgesic effects without systemic drug exposure.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To ensure double-blind conditions, all syringes are prepared and numbered by an independent laboratory technician who is not involved in the experiment. Both the participants and the experimenter are blinded to the injected substance (e.g., Flupirtine, placebo, or capsaicin combinations). Due to technical limitations, blinding of the experimenter to the temperature of injected fluid is not possible; therefore, the room-temperature injection in the heat condition is single-blind. Familiarization injections are administered unblinded for safety and tolerability assessment. Blinding is maintained until the end of each subject's participation. Randomization sequences are generated and stored separately and are only accessible to unblinded personnel in case of emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Capsaicin Sequence A (Experimental): Participants receive six intradermal injections in the following order:
  1. Capsaicin 7.6 ng
  2. Capsaicin + Flupirtine 0.5 µg
  3. Capsaicin + Flupirtine 1.2 µg
  4. Capsaicin + Flupirtine 3.0 µg
  5. Capsaicin + Flupirtine 7.6 µg
  6. Placebo (SIF only) Pain is rated every 5 seconds. Each injection is blinded and separated by ≥3 cm.
  Interventions: Drug: Capsaicin only (7.6 ng); Drug: Capsaicin + Flupirtine 0.5 µg; Drug: Capsaicin + Flupirtine 1.2 µg; Drug: Capsaicin + Flupirtine 3.0 µg; Drug: Capsaicin + Flupirtine 7.6 µg; Drug: Placebo (SIF only, no capsaicin or Flupirtine)
- Capsaicin Sequence B (Experimental): Same interventions as Sequence A but in a different order according to Williams design.
  Interventions: Drug: Capsaicin only (7.6 ng); Drug: Capsaicin + Flupirtine 0.5 µg; Drug: Capsaicin + Flupirtine 1.2 µg; Drug: Capsaicin + Flupirtine 3.0 µg; Drug: Capsaicin + Flupirtine 7.6 µg; Drug: Placebo (SIF only, no capsaicin or Flupirtine)
- Capsaicin Sequence C (Experimental): Same interventions as Sequence A but in a different order according to Williams design.
  Interventions: Drug: Capsaicin only (7.6 ng); Drug: Capsaicin + Flupirtine 0.5 µg; Drug: Capsaicin + Flupirtine 1.2 µg; Drug: Capsaicin + Flupirtine 3.0 µg; Drug: Capsaicin + Flupirtine 7.6 µg; Drug: Placebo (SIF only, no capsaicin or Flupirtine)
- Capsaicin Sequence D (Experimental): Same interventions as Sequence A but in a different randomized order according to Williams design.
  Interventions: Drug: Capsaicin only (7.6 ng); Drug: Capsaicin + Flupirtine 0.5 µg; Drug: Capsaicin + Flupirtine 1.2 µg; Drug: Capsaicin + Flupirtine 3.0 µg; Drug: Capsaicin + Flupirtine 7.6 µg; Drug: Placebo (SIF only, no capsaicin or Flupirtine)
- Capsaicin Sequence E (Experimental): Same interventions as Sequence A but in a different order according to Williams design
  Interventions: Drug: Capsaicin only (7.6 ng); Drug: Capsaicin + Flupirtine 0.5 µg; Drug: Capsaicin + Flupirtine 1.2 µg; Drug: Capsaicin + Flupirtine 3.0 µg; Drug: Capsaicin + Flupirtine 7.6 µg; Drug: Placebo (SIF only, no capsaicin or Flupirtine)
- Capsaicin Sequence F (Experimental): Same interventions as Sequence A but in a different order according to Williams design.
  Interventions: Drug: Capsaicin only (7.6 ng); Drug: Capsaicin + Flupirtine 0.5 µg; Drug: Capsaicin + Flupirtine 1.2 µg; Drug: Capsaicin + Flupirtine 3.0 µg; Drug: Capsaicin + Flupirtine 7.6 µg; Drug: Placebo (SIF only, no capsaicin or Flupirtine)
- Heat Sequence A (Experimental): Participants receive three slow increasingly warm intradermal injections in the following order:
  1. Room temperature SIF (control)
  2. Heated SIF (placebo)
  3. Heated SIF + Flupirtine 124 µg Injections are randomized using a Williams design. Pain is rated every 5 seconds until 6 consecutive zeros.
  Interventions: Drug: Room Temperature Injection (Control); Drug: Heated injection without Flupirtine; Drug: Heated Injection with Flupirtine 124 µg
- Heat Sequence B (Experimental): Same injections as Heat Sequence A, administered in a different order according to Williams design.
  Interventions: Drug: Room Temperature Injection (Control); Drug: Heated injection without Flupirtine; Drug: Heated Injection with Flupirtine 124 µg
- Heat Sequence C (Experimental): Same injections as Heat Sequence A, administered in a different order according to Williams design.
  Interventions: Drug: Room Temperature Injection (Control); Drug: Heated injection without Flupirtine; Drug: Heated Injection with Flupirtine 124 µg
- Heat Sequence D (Experimental): Same injections as Heat Sequence A, administered in a different order according to Williams design.
  Interventions: Drug: Room Temperature Injection (Control); Drug: Heated injection without Flupirtine; Drug: Heated Injection with Flupirtine 124 µg
- Heat Sequence E (Experimental): Same injections as Heat Sequence A, administered in a different order according to Williams design.
  Interventions: Drug: Room Temperature Injection (Control); Drug: Heated injection without Flupirtine; Drug: Heated Injection with Flupirtine 124 µg
- Heat Sequence F (Experimental): Same injections as Heat Sequence A, administered in a different order according to Williams design.
  Interventions: Drug: Room Temperature Injection (Control); Drug: Heated injection without Flupirtine; Drug: Heated Injection with Flupirtine 124 µg

INTERVENTIONS:
Drug: Capsaicin only (7.6 ng) — Intradermal injection of 7.6 ng capsaicin (0.5 µM, 50 µL) in synthetic interstitial fluid (SIF) without Flupirtine. Used to induce experimental burning pain in the skin.
  Arms: Capsaicin Sequence A; Capsaicin Sequence B; Capsaicin Sequence C; Capsaicin Sequence D; Capsaicin Sequence E; Capsaicin Sequence F
Drug: Capsaicin + Flupirtine 0.5 µg — Intradermal co-injection of 7.6 ng capsaicin (0.5 µM) and 0.5 µg Flupirtine in 50 µL SIF. Used to assess local analgesic effect of very low-dose Flupirtine on chemically induced pain.
  Arms: Capsaicin Sequence A; Capsaicin Sequence B; Capsaicin Sequence C; Capsaicin Sequence D; Capsaicin Sequence E; Capsaicin Sequence F
Drug: Capsaicin + Flupirtine 1.2 µg — Intradermal co-injection of 7.6 ng capsaicin and 1.2 µg Flupirtine in 50 µL SIF. Part of dose-response evaluation for peripheral pain inhibition.
  Arms: Capsaicin Sequence A; Capsaicin Sequence B; Capsaicin Sequence C; Capsaicin Sequence D; Capsaicin Sequence E; Capsaicin Sequence F
Drug: Capsaicin + Flupirtine 3.0 µg — Intradermal co-injection of 7.6 ng capsaicin and 3.0 µg Flupirtine in 50 µL SIF. Intermediate dose in microdose titration series.
  Arms: Capsaicin Sequence A; Capsaicin Sequence B; Capsaicin Sequence C; Capsaicin Sequence D; Capsaicin Sequence E; Capsaicin Sequence F
Drug: Capsaicin + Flupirtine 7.6 µg — Intradermal co-injection of 7.6 ng capsaicin and 7.6 µg Flupirtine in 50 µL SIF. This is the highest Flupirtine microdose used in the capsaicin model.
  Arms: Capsaicin Sequence A; Capsaicin Sequence B; Capsaicin Sequence C; Capsaicin Sequence D; Capsaicin Sequence E; Capsaicin Sequence F
Drug: Placebo (SIF only, no capsaicin or Flupirtine) — Intradermal injection of 50 µL synthetic interstitial fluid without capsaicin or Flupirtine. Used as negative control for capsaicin-Flupirtine co-injection conditions.
  Arms: Capsaicin Sequence A; Capsaicin Sequence B; Capsaicin Sequence C; Capsaicin Sequence D; Capsaicin Sequence E; Capsaicin Sequence F
Drug: Room Temperature Injection (Control) — Intradermal slow infusion of SIF at ~23°C using a programmable pump. No capsaicin or Flupirtine included. Used as baseline control in heat model.
  Arms: Heat Sequence A; Heat Sequence B; Heat Sequence C; Heat Sequence D; Heat Sequence E; Heat Sequence F
Drug: Heated injection without Flupirtine — Intradermal slow infusion of synthetic interstitial fluid preheated up to ~52°C. No Flupirtine included. Used to induce thermal pain in human skin.
  Arms: Heat Sequence A; Heat Sequence B; Heat Sequence C; Heat Sequence D; Heat Sequence E; Heat Sequence F
Drug: Heated Injection with Flupirtine 124 µg — Intradermal slow infusion of synthetic interstitial fluid up to ~52°C containing 124 µg Flupirtine. Used to test local analgesic effect of high-dose Flupirtine in heat pain model.
  Arms: Heat Sequence A; Heat Sequence B; Heat Sequence C; Heat Sequence D; Heat Sequence E; Heat Sequence F

SUMMARY:
The goal of this clinical trial is to learn if the drug Flupirtine can safely lower pain when used in tiny amounts directly in the skin. The study will test whether Flupirtine works by activating specific nerve channels in the skin called KV7 potassium channels. These channels help control how pain signals travel to the brain.

The main questions the study aims to answer are:

* Does Flupirtine lower pain caused by capsaicin, the active ingredient in chili peppers?
* Does Flupirtine lower pain caused by heat?

Researchers will compare Flupirtine to a placebo (a look-alike injection that does not contain any drug) to see if Flupirtine lowers pain better than the placebo.

Participants will:

* Receive tiny skin injections that contain either Flupirtine, capsaicin, heat, or placebo
* Rate their pain on a scale from 0 (no pain) to 100 (worst pain imaginable)
* Complete all study procedures during one visit that lasts about 1 hour

Only a small amount of Flupirtine will be used in this study-less than 1/800 of the usual dose. The drug is injected into the skin, not taken by mouth. Because of this, the risk of side effects is extremely low.

This study includes healthy adults between the ages of 18 and 70. It does not include people who are pregnant, taking medications, or who have skin or nerve problems.

The goal is to find out if Flupirtine can be used in the future to treat pain in a new way-by working directly in the skin and not in the brain. This could help avoid side effects like tiredness or dizziness.

The study is sponsored by the Medical University of Vienna and follows all safety and ethical rules.

DETAILED DESCRIPTION:
This randomized, placebo-controlled crossover clinical trial investigates whether a very small (microdose) amount of the drug Flupirtine, when injected directly into the skin, can reduce pain caused by chemical and heat-based stimuli. The research is based on the hypothesis that activating KV7 potassium channels in peripheral sensory nerves can lower pain without involving the central nervous system (brain and spinal cord), potentially offering a new class of non-opioid analgesics with fewer side effects.

Background and Rationale

Pain is the leading reason why people seek medical care. While several types of pain medications exist-such as non-opioid and opioid analgesics, antidepressants, anticonvulsants, and local anesthetics-many have limitations due to side effects, addiction risks, or limited effectiveness in certain pain types. New strategies for safe, targeted pain relief are urgently needed.

Recent research highlights KV7 channels, a group of voltage-gated potassium channels, as promising targets for pain modulation. These channels are expressed in peripheral sensory neurons, including nociceptors in the skin. When activated, they make it less likely for the neuron to send pain signals to the brain. Preclinical studies in animals have shown that activating these channels-particularly the KV7.2/7.3 subtypes-can reduce pain.

Flupirtine, a previously approved non-opioid analgesic, is known to activate KV7 channels. Although it was withdrawn from the market due to rare cases of liver toxicity after long-term, high-dose systemic use, its mechanism of action remains of high scientific interest. Importantly, prior studies suggest that Flupirtine's pain-relieving effects may occur, at least in part, through peripheral activation of KV7 channels.

In this study, Flupirtine is used at doses over 800 times lower than those associated with any systemic toxicity, and is applied locally into the skin to restrict its action to the peripheral nervous system. This "microdosing" strategy is intended to eliminate systemic exposure while retaining local analgesic potential.

Study Objectives

Primary Objective 1:

To test whether pain caused by intradermal injection of 7.6 ng capsaicin (a TRPV1 agonist) is reduced by co-injection of 7.6 µg Flupirtine.

Primary Objective 2:

To test whether pain caused by a slow, intradermal injection of heated fluid (up to ~52°C) is reduced by co-injection of 124 µg Flupirtine.

Secondary Objectives:

* To explore dose-response relationships for lower doses of Flupirtine (0.5 µg, 1.2 µg, 3.0 µg) in the capsaicin pain model.
* To observe pain patterns across all injection types in a within-subjects crossover design.

Study Design

This is a two-part, single-visit, crossover trial in healthy adult volunteers. The study uses a Williams design to balance for injection sequence and period effects.

Each participant undergoes:

* 7 intradermal bolus injections: 1 unblinded familiarization with capsaicin, followed by 6 blinded, randomized injections containing capsaicin ± varying doses of Flupirtine or placebo.
* 4 intradermal slow infusions: 1 unblinded familiarization with room-temperature fluid, followed by 3 blinded, randomized heat infusions with or without Flupirtine.

Each injection site is separated by at least 3 cm on alternating volar forearms. All injections are performed under sterile conditions.

Pain is rated by participants every 5 seconds on a 0-100 numerical scale. Pain ratings continue until the participant reports zero pain for 30 seconds. Pain Area Under the Curve (Pain AUC) is calculated using the trapezoidal rule and serves as the primary outcome.

The total Flupirtine dose per subject across all injections is 136.3 µg, which is less than 0.14 mg, well below known toxicity thresholds. The vehicle for injection is synthetic interstitial fluid with 0.5% DMSO and 0.1% polysorbate 80.

Safety Considerations

Flupirtine's known risk profile includes liver toxicity only after prolonged, high-dose systemic use (200-600 mg daily for >14 days). This study uses:

* A single dose of <0.14 mg
* Local intradermal administration, not systemic
* No follow-up dosing

These differences make hepatotoxicity highly unlikely. In addition, no local tissue toxicity is expected, as previous injectable formulations (e.g., Katadolon inject) contained over 100 mg per 3 mL with no reported injection-site damage.

The other injected agent, capsaicin, is widely used in experimental pain research. The dose (7.6 ng in 50 µL) is much lower than in similar studies and causes only brief burning pain with no lasting effects.

Adverse events (AEs) and serious adverse events (SAEs) will be recorded. These may include:

* Mild local skin reactions (e.g., redness, itch)
* Injection site bleeding
* Rare allergic reactions

No follow-up visits are planned, but participants are informed to report any delayed symptoms.

Statistical Analysis

Primary analyses will be performed on the per-protocol set to ensure integrity of the crossover design. Supplementary intention-to-treat analyses will also be performed.

Statistical models include:

* Linear mixed models with injection type (fixed), injection period (fixed), and subject (random)
* Covariate adjustment for insertion pain
* No multiplicity correction, as both objectives are treated as independent

Sample size calculations are based on prior published data (Heber et al. 2019; unpublished heat data). A total of 32 participants will be recruited to allow for 5% dropout and balanced sex representation.

Implications and Future Directions

If successful, this study could support the development of new peripherally acting pain medications based on KV7 activation. Such drugs might avoid central nervous system side effects (like sedation or dizziness) and could represent an important alternative or supplement to current pain therapies-especially for localized inflammatory or neuropathic pain.

Furthermore, a better understanding of peripheral pain pathways could guide drug development that avoids opioid use and its associated risks.

Study Location

All procedures take place at the Department of Anesthesia, Intensive Care Medicine, and Pain Medicine at the Medical University of Vienna.

Ethics and Registration

The study has been reviewed and approved by the local Ethics Committee. It is conducted in accordance with the Declaration of Helsinki, Good Clinical Practice (GCP), and GDPR regulations.

Participants receive full information and provide written informed consent before taking part. Participation is voluntary, and withdrawal is possible at any time without giving a reason.

Results will be submitted for publication in a peer-reviewed journal and presented at relevant scientific conferences. Identifiable data will not be disclosed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Full legal capacity To ensure an equal number of each sex in the study population, only volunteers of one sex will be included as soon as the number of subjects with the other sex has reached half of the calculated sample size.

Exclusion Criteria:

* Participant of another study, ongoing or within the last 4 weeks
* Medication intake (except contraception) or drug abuse
* Female subjects: Positive pregnancy test or breastfeeding
* Body temperature above 38°C, diagnostically verified
* Known allergic diseases, in particular asthmatic disorders and skin diseases
* Sensory deficit, skin disease or hematoma of unknown origin in examination of the test site

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity over time (area under the curve, AUC) after intradermal capsaicin or heat stimulus ± Flupirtine | Immediately post-injection, up to 3 minutes on Day 1
  Pain is rated every 5 seconds using a numerical rating scale from 0 (no pain) to 100 (worst imaginable pain). Ratings continue until the participant reports zero pain for 30 consecutive seconds. For each injection, the area under the curve (AUC) of pain intensity over time is calculated. The primary outcome is the difference in pain AUC between Flupirtine-treated and placebo-treated conditions in both the capsaicin and heat models.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including pain ratings, time-stamped injection responses, and basic demographics (age, sex), will be shared after publication of the primary results. Only data used in the main publication and relevant supplementary analyses will be included.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be made available at the time of publication of the primary results article, as a supplementary file.
Access Criteria: All individuals who have access to the published article will be able to access the individual participant data (IPD) and supporting information as supplementary material. No special request or data use agreement is required.

REFERENCES:
- [Background] Heber S, Resch F, Ciotu CI, Gleiss A, Heber UM, Macher-Beer A, Bhuiyan S, Gold-Binder M, Kain R, Sator S, Fischer MJM. Human heat sensation: A randomized crossover trial. Sci Adv. 2024 Sep 6;10(36):eado3498. doi: 10.1126/sciadv.ado3498. Epub 2024 Sep 4. PMID 39231217
- [Background] Heber S, Gold-Binder M, Ciotu CI, Witek M, Ninidze N, Kress HG, Fischer MJM. A Human TRPA1-Specific Pain Model. J Neurosci. 2019 May 15;39(20):3845-3855. doi: 10.1523/JNEUROSCI.3048-18.2019. Epub 2019 Mar 12. PMID 30862667
- [Background] Heber S, Ciotu CI, Hartner G, Gold-Binder M, Ninidze N, Gleiss A, Kress HG, Fischer MJM. TRPV1 antagonist BCTC inhibits pH 6.0-induced pain in human skin. Pain. 2020 Jul;161(7):1532-1541. doi: 10.1097/j.pain.0000000000001848. PMID 32107360